CLINICAL TRIAL: NCT05237492
Title: The Influence of Tramadol on Platelet Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1
Record Dates: First submitted 2021-12-18; First posted 2022-02-14 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Drug Toxicity; Platelet Dysfunction; Clotting Disorder
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Hemostatic Disorders | interventions — Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- procoagulant effect on platelet function (Experimental): LTA platelet function measurement on whole blood with addition of tramadol, demonstration of a dose-response relationship and determination of the effect of combination with other drugs.
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Tramadol — Blood samples will be drawn from 15 patients. Tramadol will be added to all this samples in-vitro and its influence on platelets´ function will be measured.

SUMMARY:
The aim of this ex-vivo study is to quantify the effect of tramadol on platelet aggregation.

DETAILED DESCRIPTION:
The aim of this study is to quantify the effect of tramadol on platelet aggregation. To this end, the effect of tramadol on platelet function will be demonstrated in an ex-vivo study using optical aggregometry (LTA) on whole blood of 15 patients.

The main objective variable is to use platelet function assays (LTA) as well as thrombelastography (TEG) to determine this effect on platelet function.

The null hypothesis of this study is that tramadol does not affect platelet aggregation in healthy patients.

In addition, two further questions will be addressed:

* using a titration series, to attempt to plot a dose/response curve of the effect of tramadol on platelet function.
* tramadol is often administered together with other drugs such as NSAIDs (ibuprofen), novalgin, SSRIs or other opioids such as morphine or in the surgical setting fentanyl and remifentanil. A series of studies will be conducted to determine whether these combinations alter the effect of tramadol on platelet function.

ELIGIBILITY:
Inclusion Criteria:

* 18y and older, healthy volunteers

Exclusion Criteria:

* Age < 18 years
* Pregnant women
* History of addiction (especially opiate abuse)
* Pre-existing general addictive disease
* Ongoing pain therapy with opiates
* Taking antidepressants (SNRI, SSRI)
* History of thrombocytopathy or coagulation disorders
* Therapy with drugs that influence thrombocyte function (ASS, clopidogrel, prasugrel, ticagrelor or similar)
* Known intolerance to opiates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Procoagulant effect on platelet function demonstrated by optical aggregometry (LTA) on whole blood. | up to 4 hours
  The effect of tramadol on platelet function will be demonstrated in an ex-vivo study using optical aggregometry (LTA) on whole blood of 15 patients. The study team expects a noticeable procoagulant effect due to the increase in serotonin in the synaptic cleft in the LTA platelet function measurement by ADP, both in AUC and graphically represented as a curve.

SECONDARY OUTCOMES:
Dose/ Response - Curve | up to 4 hours
  The study team will use a titration series, to attempt to plot a dose/response curve of the effect of tramadol on platelets´ function. This question is examined on half of the blood samples (7).
Combinations with Tramadol and other drugs and their procoagulant effect on platelet function demonstrated by optical aggregometry (LTA) on whole blood. | up to 4 hours
  Tramadol is often administered together with other drugs such as NSAIDs (ibuprofen), novalgin, SSRIs or other opioids such as morphine or in the surgical setting fentanyl and remifentanil. A series of studies will be conducted to determine whether these combinations alter the effect of tramadol on platelet function. This question will be examined on the other half of the whole blood samples (7) and measured in the LTA platelet function measurement by ADP, both in AUC and graphically represented as a curve.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Zoidl, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Dept. of Anaesthesiology and Intensive Care Medicine, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: CSR, Analytic Code
Time Frame: As soon as results are published, ca early 2023